CLINICAL TRIAL: NCT00359177
Title: An Open-Label, Non-Randomized, Pharmacokinetic and Safety Study of Multiple Oral Doses of GW679769 in Subjects With Hepatic Impairment
Brief Title: Observational Study Evaluating The Processing Or Breakdown Of GW679769 In Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKT102785
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Vomiting
Keywords: emesis liver problems hepatic impairment GW679769
MeSH Terms: conditions — Vomiting | interventions — casopitant

ARMS (2):
- Healthy subjects receiving GW679769 (Experimental): Healthy Subjects will receive single 100 milligram (mg) oral doses of GW679769 for five consecutive days.
  Interventions: Drug: GW679769
- Subjects with hepatic impairment receiving GW679769 (Experimental): Subjects with hepatic impairment will receive single 100 mg oral doses of GW679769 for five consecutive days.
  Interventions: Drug: GW679769

INTERVENTIONS:
Drug: GW679769 — GW679769 will be available in dose strength of 50 mg tablets. Subjects will receive two tablets of 50 mg orally once daily in the morning

SUMMARY:
The purpose of the study is to evaluate how subjects with mild or moderate liver problems process or breakdown the study drug GW679769 in their bodies as compared to healthy subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy or have mild or moderate hepatic impairment
* Females: Non-childbearing (hysterectomy, bilateral oophorectomy, post-menopausal), childbearing (negative pregnancy test, abstinence, double-barrier contraception, vasectomized partner)
* Negative for Hepatitis B and C(healthy subjects)
* Negative drug, alcohol and HIV tests

Exclusion criteria:

* Fluctuating or rapidly deteriorating hepatic function or abnormal kidney function
* Encephalopathy
* Active peptic ulcer disease
* Drug or alcohol abuse
* Pregnant or lactating
* Esophageal bleeding
* Heart failure
* Infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2006-10-12 (Actual); Study Completion 2006-10-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) of single oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for pharmacokinetics (PK) analysis will be collected at the indicated time points. AUC will be calculated from plasma GW679769 concentration.
AUC of multiple oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. AUC will be calculated from plasma GW679769 concentration.
AUC of single oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. AUC will be calculated from plasma GW679769 concentration.
AUC of multiple oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. AUC will be calculated from plasma GW679769 concentration.
Maximum observed concentration (Cmax) of single oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GW679769 concentration.
Cmax of multiple oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GW679769 concentration.
Cmax of single oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GW679769 concentration.
Cmax of multiple oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GW679769 concentration.
AUC of single oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. AUC will be calculated from plasma GSK525060 concentration.
AUC of multiple oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. AUC will be calculated from plasma GSK525060 concentration.
AUC of single oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. AUC will be calculated from plasma GSK525060 concentration.
AUC of multiple oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. AUC will be calculated from plasma GSK525060 concentration.
Cmax of single oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GSK525060 concentration.
Cmax of multiple oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GSK525060 concentration
Cmax of single oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GSK525060 concentration.
Cmax of multiple oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. Cmax will be calculated from plasma GSK525060 concentration.

OTHER OUTCOMES:
Time to maximum observed concentration (tmax) of single oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GW679769 concentration-time data.
tmax of multiple oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GW679769 concentration-time data.
tmax of single oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GW679769 concentration-time data.
tmax of multiple oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GW679769 concentration-time data.
tmax of single oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GSK525060 concentration-time data.
tmax of multiple oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GSK525060 concentration-time data.
tmax of single oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GSK525060 concentration-time data.
tmax of multiple oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. tmax will be calculated from plasma GSK525060 concentration-time data.
Terminal half-life (t1/2) of single oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GW679769 concentration-time data.
t1/2 of multiple oral dose of GW679769 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GW679769 concentration-time data.
t1/2 of single oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GW679769 concentration-time data.
t1/2 of single oral dose of GW679769 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GW679769 concentration-time data.
t1/2 of single oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GSK525060 concentration-time data.
t1/2 of multiple oral dose of GSK525060 in healthy subjects | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GSK525060 concentration-time data.
t1/2 of single oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GSK525060 concentration-time data
t1/2 of multiple oral dose of GSK525060 in subjects with mild and moderate hepatic impairment | Day 1 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours, Pre-dose (Day 3 and 4), Day 5 Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours
  Blood samples for PK analysis will be collected at the indicated time points. t1/2 will be calculated from plasma GSK525060 concentration-time data
Percentage of unbound GW679769 in healthy subjects receiving single oral dose of GW679769 | 1, 2, 4 and 24 hours post-dose on Day 1
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GW679769 will be calculated from plasma GW679769 concentration-time data.
Percentage of unbound GW679769 in healthy subjects receiving multiple oral dose of GW679769 | 1, 2, 4 and 24 hours post-dose on Day 1. Day 5, Pre-dose, 1, 2, 4, 24 hours post-dose
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GW679769 will be calculated from plasma GW679769 concentration-time data
Percentage of unbound GW679769 in subjects with mild and moderate hepatic impairment receiving single oral dose of GW679769 | 1, 2, 4 and 24 hours post-dose on Day 1
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GW679769 will be calculated from plasma GW679769 concentration-time data.
Percentage of unbound GW679769 in subjects with mild and moderate hepatic impairment receiving multiple oral dose of GW679769 | 1, 2, 4 and 24 hours post-dose on Day 1. Day 5, Pre-dose, 1, 2, 4, 24 hours post-dose
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GW679769 will be calculated from plasma GW679769 concentration-time data.
Percentage of unbound GSK525060 in healthy subjects receiving single oral dose of GSK525060 | 1, 2, 4 and 24 hours post-dose on Day 1
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GSK525060 will be calculated from plasma GSK525060 concentration-time data.
Percentage of unbound GSK525060 in healthy subjects receiving multiple oral dose of GSK525060 | 1, 2, 4 and 24 hours post-dose on Day 1. Day 5, Pre-dose, 1, 2, 4, 24 hours post-dose
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GSK525060 will be calculated from plasma GSK525060 concentration-time data.
Percentage of unbound GSK525060 in subjects with mild and moderate hepatic impairment receiving single oral dose of GSK525060 | 1, 2, 4 and 24 hours post-dose on Day 1
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GSK525060 will be calculated from plasma GSK525060 concentration-time data.
Percentage of unbound GSK525060 in subjects with mild and moderate hepatic impairment receiving multiple oral dose of GSK525060 | 1, 2, 4 and 24 hours post-dose on Day 1. Day 5, Pre-dose, 1, 2, 4, 24 hours post-dose
  Blood samples for PK analysis will be collected at the indicated time points. Percentage of unbound GSK525060 will be calculated from plasma GSK525060 concentration-time data.
Number of subjects with Adverse events (AE) and Serious AEs (SAE) | Up to Day 22
  An AE is any untoward medical occurrence in a clinical study subject, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that at any dose may result in death, is life-threatening, may require hospitalization or prolongation of existing hospitalization, result in persistent disability/incapacity, or may led to any congenital anomaly or birth defect
Number of subjects with abnormal systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Up to Day 22
  Blood pressure measurement will be assessed in supine and resting position.
Number of subjects with abnormal heart rate | Up to Day 22
  Blood pressure measurement will be assessed in supine and resting position.
Number of subjects with abnormal hematology parameters | Up to Day 22
  Laboratory assessment for hematology parameters will include hemoglobin, hematocrit, red blood cell count (RBC), platelet count, white blood cell count (WBC), neutrophil count, lymphocyte count, monocyte count, eosinophil count, basophil count, prothrombin time (PT), and International Normalized Ratio (INR)
Number of subjects with abnormal clinical chemistry parameters | Up to Day 22
  Laboratory assessment for clinical chemistry parameters sodium, potassium, chloride, total Carbon dioxide, calcium, glucose (fasting), phosphorous (inorganic), protein (total), albumin, gamma-glutamyl-transferase (GGT), bilirubin (total), alkaline Phosphatase, lactic dehydrogenase (LDH), aspartate aminotransferase (AST; Serum glutamic oxaloacetic transaminase), alanine aminotransferase (ALT; Serum glutamic pyruvic transaminase), creatinine, blood Urea Nitrogen, uric Acid, creatine Phosphokinase (CPK), and ammonia
Number of subjects with abnormal urinalysis | Up to Day 22
  Laboratory assessment for urinalysis parameters pH, specific gravity, glucose, protein, ketones, and blood

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study NKT102785 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/NKT102785?search=study&search_terms=NKT102785#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: NKT102785 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKT102785 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKT102785 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKT102785 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKT102785 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKT102785 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKT102785 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register